CLINICAL TRIAL: NCT01644006
Title: Telemedical Support in Prehospital Emergency Care of Acute Coronary Syndromes
Brief Title: Telemedical Support in Prehospital Emergency Care of Acute Coronary Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: RWTH Aachen University (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 005-1003-0034-1; PtJ-Az.: z0909im002b (Other Grant/Funding Number: PTJ)
Record Dates: First submitted 2012-07-12; First posted 2012-07-18 (Estimated); Last update posted 2015-09-22 (Estimated); Status verified 2015-09

CONDITIONS: Acute Coronary Syndrome
Keywords: acute coronary syndrome; telemedicine; teleconsultation; emergency medical service
MeSH Terms: conditions — Acute Coronary Syndrome | interventions — Remote Consultation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Device: Teleconsultation (Experimental): In cases of suspected acute coronary syndrome (including STEMI), if patients give informed consent the paramedics can use this system to contact a so called "tele-EMS physician" with audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. Also 12-lead-ECGs can be transmitted to the tele-EMS physician. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, ECG diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene.
  The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.
  Interventions: Procedure: Teleconsultation
- Historical Matched Pairs (No Intervention): Historical matched pairs were searched from local protocols. During this phase no teleconsultation system was existent.

INTERVENTIONS:
Procedure: Teleconsultation — Teleconsultation of an EMS physician to support the paramedics in acute coronary syndromes
  Arms: Device: Teleconsultation

SUMMARY:
The aim of the study is to investigate the quality of prehospital emergency care in acute coronary syndromes, when paramedics are supported telemedically by an EMS physician.

DETAILED DESCRIPTION:
Six ambulances from five different Emergency Medical Service (EMS) districts are equipped with a portable telemedicine system. In cases of suspected acute coronary syndrome (including STEMI), the paramedics can use this system to contact a so called "tele-EMS physician" after consent of the patient is obtained. The tele-EMS physician has an audio-connection to the EMS team and receives vital parameters (e.g., ECG, pulse oximetry, non-invasive blood pressure) in real-time. Also 12-lead-ECGs can transmitted to the tele-EMS physician. The transmission of still pictures - taken with a smartphone - and video streaming from the inside of the ambulance can be carried out, if meaningful. The tele-EMS physician supports the EMS team in obtaining all relevant medical history, ECG diagnosis, general diagnosis and can delegate the application of medications. This can be carried out to bridge the time to the arrival of an EMS physician or in less severe cases without an EMS physician on-scene.

The quality of prehospital care and the possible influences on the initial inhospital phase should be investigated and compared with regular EMS.

ELIGIBILITY:
Inclusion Criteria:

* Suspected acute coronary syndrome
* Verbal consent for teleconsultation obtained or patient is not able to consent due to the severity of the emergency

Exclusion Criteria:

* Patient refuses consent to teleconsultation
* No suspected acute coronary syndrome

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2012-08; Primary Completion 2013-07 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Quality of prehospital care | average 1 hour
  Analysis of the quality of the prehospital care on the basis of published guidelines for ACS / STEMI

SECONDARY OUTCOMES:
Inhospital time intervals in STEMI | up to 12 hours
  contact to balloon time, arrival to balloon time
Rate of secondary transfer for PCI | up to 7 days
  Rate of secondary transfer to a different facility for PCI
Troponin-Level | 24 hours
  Severity of infarction measured with level of Troponin
Conducted procedures and medications (paramedics) | average 1 hour
  Amount of guidelines based procedures and medications carried out by paramedics prior to the contact with a physician.
prehospital time intervals | average 1 hour
  on-scene time, contact (EMS) to hospital arrival time, transport time

CONTACTS AND LOCATIONS:
Overall Officials: Rolf Rossaint, Prof. Dr., Study Chair — University Hospital Aachen, Germany, Department of Anesthesiology; Jörg C Brokmann, Dr., Principal Investigator — University Hospital Aachen, Germany, Emergency Department
Locations (1):
- University Hospital Aachen, Aachen, Germany

REFERENCES:
- [Derived] Brokmann JC, Conrad C, Rossaint R, Bergrath S, Beckers SK, Tamm M, Czaplik M, Hirsch F. Treatment of Acute Coronary Syndrome by Telemedically Supported Paramedics Compared With Physician-Based Treatment: A Prospective, Interventional, Multicenter Trial. J Med Internet Res. 2016 Dec 1;18(12):e314. doi: 10.2196/jmir.6358. PMID 27908843